CLINICAL TRIAL: NCT00871884
Title: The Role of Anxiety Sensitivity in the Maintenance of Chronic Post Concussion Symptoms
Brief Title: Evaluation of Two Treatments for Chronic Post Concussion Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor enrollment, low recruitment.
Sponsor: Simon Fraser University (Other)
Responsible Party: Principal Investigator, Kevin Whitfield, Research Coordinator, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1234567
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Post Concussion Syndrome; Head Injury
Keywords: Post Concussion Syndrome; Cognitive Behavioral Therapy; Anxiety Sensitivity; Mild Head Injury; Psychotherapy; Chronic Post Concussion Symptoms
MeSH Terms: conditions — Post-Concussion Syndrome; Craniocerebral Trauma | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment As Usual (Active Comparator)
  Interventions: Behavioral: Psychoeducation; Behavioral: Relaxation Training
- Experimental (Experimental)
  Interventions: Behavioral: Psychoeducation; Behavioral: Relaxation Training; Behavioral: Interoceptive Exposure

INTERVENTIONS:
Behavioral: Psychoeducation — Education about the common prognostic considerations, normal symptoms experienced and etiology of symptoms following mild head injury. Includes some basic suggestions surrounding methods to diminish the impact of symptoms on one's life.
Behavioral: Relaxation Training — Includes Progressive Muscle Relaxation, Guided Visualization, and various other relaxation techniques to induce deep relaxation.
Behavioral: Interoceptive Exposure — Includes a variety of exercises used to elicit somatic sensations which may be feared by the participant, in an attempt to extinguish or lessen the fear reaction to these sensations.
  Arms: Experimental

SUMMARY:
This study is designed to investigate factors that are associated with prolonged recovery from mild head injury. The investigators are particularly interested in defining the impact of anxiety related variables, such as health anxiety and anxiety sensitivity in the maintenance of symptoms.

A further goal of the study is the evaluation of two treatment methods that have been proposed to be effective in reducing the impact of post concussion symptoms. The investigators hypothesize that a treatment which is directly focused on changing these anxiety related variables will be more effective than one that does not.

ELIGIBILITY:
Inclusion Criteria:

* Mild Head Injury at least 3 months prior to treatment
* age 19 to 65 years
* grade 12 education
* proficiency with English language

Exclusion Criteria:

* Current Litigation

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Post Concussion Symptom Checklist | 0 weeks, 2 weeks, 4 weeks, 6 weeks

SECONDARY OUTCOMES:
Anxiety Sensitivity Index | 0 weeks, 2 weeks, 4 weeks, 6 weeks
State Trait Anxiety Inventory | 0 weeks, 2 weeks, 4 weeks, 6 weeks
Zung Self Rated Depression Scale | 0 weeks, 2 weeks, 4 weeks, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Whitfield, M.A., Principal Investigator — Human Neuropsychology Laboratory, Department of Psychology, Simon Fraser University; Allen E Thornton, Ph.D., Study Director — Human Neuropsychology Laboratory, Department of Psychology, Simon Fraser University; Alex P Chapman, Ph.D., Study Director — Department of Psychology, Simon fraser University; David Cox, Ph.D., Study Director — Department of Psychology, Simon Fraser University
Locations (1):
- Clinical Psychology Centre, Simon Fraser University, Burnaby, British Columbia, Canada

REFERENCES:
- See also: study recruitment homepage — http://sfuconcussionstudy.googlepages.com/home